CLINICAL TRIAL: NCT05107037
Title: A Phase I Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of TQ-B3234 Capsules in Chinese Patients With Type I Neurofibromatosis (Neurofibromatosis and Malignant Peripheral Nerve Sheath Tumors)
Brief Title: A Clinical Trial to Evaluate the Tolerability and Pharmacokinetics of TQ-B3234 in Patients With Type I Neurofibromatosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3234-I-02
Record Dates: First submitted 2021-09-03; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-06

CONDITIONS: Type I Neurofibromatosis
MeSH Terms: conditions — Neurofibromatoses

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3234 capsule (Experimental): In the dose escalation phase, enrolled subjects first received a single dose on an empty stomach for a 3-day observation period. If Dose limiting toxicity (DLT) did not occur, continuous multiple doses were continued, once a day on an empty stomach for a treatment cycle of 28 days.
  After the dose escalation phase was completed, cohort extension studies were conducted according to the identified phase ii clinical recommended doses.type I neurofibromatosis （NF1） patients and malignant peripheral nerve sheath tumors （MPNST） patients were selected.
  Interventions: Drug: TQ-B3234 capsule

INTERVENTIONS:
Drug: TQ-B3234 capsule — TQ-B3234 is an anti-tumor molecular targeted drug, which is a selective Mitogen-activated protein kinase kinase（MEK）1/2 inhibitor

SUMMARY:
This study is a Phase I clinical trial to evaluate the tolerability and pharmacokinetics of TQ-B3234 capsules in Chinese subjects associated with neurofibromatosis type I (neurofibroma and peripheral malignant neurilemmoma).

Two study phases were designed, including (1) dose escalation and (2) cohort expansion.

The purpose of this study was to evaluate the tolerance, pharmacokinetic characteristics, efficacy and safety of TQ-B3234 capsule, and to explore the therapeutic biomarkers related to this product.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily join the study, Sign the informed consent form;
2. Aged: [18~75] years old (when signing informed consent); Eastern cooperative oncology group performance Status（ECOG PS )score: ≤2 points; patients with malignant peripheral nerve sheath tumors （MPNST）are expected to survive ≥12 weeks;
3. NF1 patients (including patients with malignant peripheral nerve sheath tumor (MPNST)) who are judged by the investigator as incomplete surgical resection, require systemic treatment, and have measurable lesions;

Note: NF1 diagnostic criteria meets at least one of the following:

1. Genetic examination confirmation: test positive for NF1 germline mutation in a CLIA-certified laboratory (positive NF1 germline mutation must be confirmed by the central laboratory of this project, or an NF1 mutation test report issued by a CLIA-certified laboratory;
2. Clinical and imaging examination confirmation: According to the clinical National Institutes of Health(NIH) consensus criteria, at least two of the following seven NF1 diagnostic criteria are met:

   1. Six or more café-au-lait macules (≥0.5cm in prepubertal patients or ≥1.5 cm in post pubertal patients)
   2. Freckling in axilla or groin
   3. ≥2 neurofibromas of any type, or ≥1 plexiform neurofibromas
   4. Optic glioma
   5. Two or more Lisch nodules
   6. A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   7. A first-degree relative with NF1

      4. Confirmed by direct measurement or according to the Response Evaluation Criteria in Solid Tumors( RECIST) 1.1 standard that there is at least one evaluable lesion;

      5. The main organs function well and meet the following standards:

1) Blood routine examination standard (no blood transfusion and no hematopoietic stimulating factor drugs used for correction within 7 days before the examination):

1. White blood cell count (WBC) ≥3.5×109/L
2. Hemoglobin (HGB) ≥90 g/L;
3. The absolute value of neutrophils (NEUT) ≥ 1.5×109/L;
4. Platelet count (PLT) ≥ 100×109/L. 2) The biochemical inspection shall meet the following standards:

a. Albumin (ALB) ≥35g/L; b. Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN), and patients with Gilbert syndrome are ≤ 2.5 times the upper limit of normal (ULN); c. Alanine-based transferase (ALT) and aspartate-based transferase (AST) ≤2.5×ULN; d. Serum creatinine (CR) ≤1.5×ULN or creatinine clearance (CCR) ≥50ml/min (application of standard Cockcroft-Gault formula); 3) The coagulation function test shall meet the following standards: International normalized ratio (INR)≤1.5×ULN (have not received anticoagulant therapy); 4) Thyroid function examination must meet the following standards: Thyroid-stimulating hormone (TSH)≤ULN; if abnormal, T3 and T4 levels should be examined, and T3 and T4 levels are normal.

5) Heart color Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.

6. Female patients of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum pregnancy test within 7 days before study entry Negative, and must be a non-lactating subject; male patients should agree to adopt avoidance measures during the study period and within 6 months after the end of the study period;

7. Patients enrolled in the second stage need to be pathologically confirmed to be enrolled in cohort 1, cohort 2 or cohort 3.

Exclusion Criteria:

1. Combined diseases and medical history:

1. Have other malignant tumors within 3 years before the first medication or is currently suffering from other malignancies The following two situations can be included in the group: other malignant tumors treated by a single operation, to achieve 5 consecutive years of disease-free survival (DFS);
2. Many factors that affect oral medications (such as dysphagia, chronic diarrhea and intestinal obstruction, etc.)
3. Unreliable toxic reactions higher than Common Terminology Criteria for Adverse Events(CTCAE) v5.0 level 1 caused by any previous treatment, excluding hair loss;
4. Received major surgical treatment or obvious traumatic injury within 28 days before the first medication;
5. Long-term unhealed wounds or fractures caused by surgery or trauma;
6. Arterial/venous thrombosis occurred within 6 months before the first medication, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
7. Have a history of psychotropic drug abuse and cannot be quit or have mental disorders
8. There are risk factors for prolonging the corrected QT interval(QTc), such as uncorrectable hypokalemia, hereditary long QT syndrome, or taking drugs that prolong the QTc interval (mainly class Ia, Ic, and III antiarrhythmic drugs) ；
9. Past or current retinal vein stenosis, retinal detachment, central retinal vein occlusion, glaucoma, grade 1 cataract, related symptoms caused by the disease are not considered as exclusion criteria;
10. Interstitial pneumonia, including clinically significant radiation pneumonia;
11. Patients with any severe and/or uncontrollable disease, including:

    1. Unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg);
    2. Suffering from grade ≥2 myocardial ischemia or myocardial infarction, arrhythmia (including male QTc ≥450 ms (male), QTc ≥470 ms (female)) and grade ≥2 congestive heart failure (New York Heart Association ( NYHA) classification, appendix 2);
    3. Active or uncontrolled serious infection (≥CTCAE v5.0 Grade 2 infection);
    4. Active hepatitis: hepatitis B reference:hepatitis b surface antigen（HBsAg） is positive, and the DNA of hepatitis B virus(HBV DNA) test value exceeds the upper limit of normal; hepatitis C reference: HCV antibody is positive, and the HCV virus titer test value exceeds the upper limit of normal; Note: Those who meet the criteria for entry, hepatitis B surface antigen-positive or core antibody-positive patients, and hepatitis C patients need to continue antiviral therapy to prevent virus activation;
    5. Renal failure requiring hemodialysis or peritoneal dialysis;
    6. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
    7. Poor diabetes control (fasting blood glucose (FBG)> 10 mmol/L);
    8. Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein quantification is confirmed to be >1.0 g;
    9. Those who suffer from epilepsy and need treatment;

       2. Tumor-related symptoms and treatment:

1) Have received surgery, chemotherapy, radiotherapy or other anti-cancer therapies within 4 weeks before the first medication (the washout period will be calculated from the end of the last treatment); 2) Have received NMPA approved Chinese patent medicines with anti-tumor indications (including compound cantharidin capsules, Kangai injections, Kanglaite capsules/injections, Aidi injections, Brucea javanica oil injections). /Capsules, Xiaoaiping Tablets/Injections, Huachansu Capsules, etc.) treatment;

3. Research and treatment related:

1. Patients who have previously received one of the following treatments:

   1. Patients who have received NF1 drug treatment within 3 months before enrollment, and the related side effects have not yet recovered to below grade 1 (except for hair loss). Note: Patients who are receiving NF1 drug treatment must recover from the acute toxicity of the current NF1 treatment to less than or equal to Grade 1 (refer to CTCAE v5.0) before entering this study;
   2. Patients Received tipifarnib, pirfenidone, peg-interferon, sorafenib or other Vascular Endothelial Growth Factor Receptor(VEGFR) inhibitor or biological treatments within 14 days before receiving study drug treatment ;
   3. Receiving strong CYP3A4 inhibitors (amprenavir, atazanavir, boceprevir, clarithromycin, cornivatan, delavirdine, diltiazem, erythromycin) within 14 days before receiving study drug treatment , Fursanavir, Indinavir, Itraconazole, Ketoconazole, Lopinavir, Mibefradil, Miconazole, Nefazodone, Nefinavir, Posaconazole, Ritonavir, saquinavir, tilarrevir, telithromycin, verapamil, voriconazole, etc.) or strong inducers (carbamazepine, felbamate, nevirapine, phenobarbital, phenytoin, Patients with primidone, rifabutin, rifampicin, rifapentine, etc.), except for external use on the skin;
2. Unable to perform Nuclear Magnetic Resonance Imaging(MRI) examination and/or there are contraindications for MRI examination, such as prosthesis, orthotics or orthodontics, which will interfere with the volume analysis of the target plexiform neurofibromas( PN) on MRI;
3. Patients who need to take more than the recommended dose of vitamin E daily;

4. Participated within 4 weeks before the first medication and used other anti-tumor clinical trial drugs or those who have not exceeded 5 drug half-lives;

5. According to the judgment of the investigator, there are situations that seriously endanger the safety of the patients or affect the completion of the research by the patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 48weeks
  If DLT occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD
Dose limiting toxicity (DLT) | Baseline up to 4 weeks
  Some drug-related toxicities occurred within 28 days of treatment
Phase II clinical recommended dose （RP2D） | Baseline up to 48 weeks
  Phase II clinical recommended dose
objective response rate（ORR） | Baseline up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Before administration, 10 , 20 , 30, 45 minuets, 1 , 2 , 4 , 6 , 10 , 24 , 48 , 72 hours after administration
  Maximum plasma drug concentration
Peak time (Tmax) | Before administration, 10 , 20 , 30, 45 minuets, 1 , 2 , 4 , 6 , 10 , 24 , 48 , 72 hours after administration
  Time to maximum plasma concentration
Clearance half-life (t1/2) | Before administration, 10 , 20 , 30, 45 minuets, 1 , 2 , 4 , 6 , 10 , 24 , 48 , 72 hours after administration
  The time required for the concentration of a drug to fall by half in a living organism
Area under plasma concentration-time Curve (AUC) | Before administration, 10 , 20 , 30, 45 minuets, 1 , 2 , 4 , 6 , 10 , 24 , 48 , 72 hours after administration
  Area under plasma concentration-time Curve
Steady state clearance half-life (t1/2, SS) | Pre-dose of day 1, day 8, day 15, day 28 on multiple dose and 10 , 20 , 30 , 45 minutes,1 , 2 , 4 , 6 , 10 , 24 hours post-dose on multiple dose of day 1 and day 28
  Steady state clearance half-life (t1/2, SS)
Plasma concentration at steady state (Cav, SS) | Pre-dose of day 1, day 8, day 15, day 28 on multiple dose and 10 , 20 , 30 , 45 minutes,1 , 2 , 4 , 6 , 10 , 24 hours post-dose on multiple dose of day 1 and day 28
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium
Area under plasma concentration-time curve at steady state (AUCss) | Pre-dose of day 1, day 8, day 15, day 28 on multiple dose and 10 , 20 , 30 , 45 minutes,1 , 2 , 4 , 6 , 10 , 24 hours post-dose on multiple dose of day 1 and day 28
  Area under plasma concentration-time curve at steady state
Coefficient of fluctuation (DF) | Pre-dose of day 1, day 8, day 15, day 28 on multiple dose and 10 , 20 , 30 , 45 minutes,1 , 2 , 4 , 6 , 10 , 24 hours post-dose on multiple dose of day 1 and day 28
  Coefficient of fluctuation
Adverse event rate | Baseline up to 96 weeks
  The occurrence of all adverse events (AE), serious adverse events (SAE) and treatment-related adverse events (TEAEs)
Progression-free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Disease Control Rate (DCR) | up to 96 weeks
  The proportion of patients whose tumor shrank or remained stable for some time, including those with complete response (CR), partial response (PR), and stable (SD).
1 year PFS rate | up to 1 year
  Rate of patients with PFS reaching 1 year among all patients
Overall survival time (OS, observed only in peripheral malignant schwannomas) | up to 5 year
  The time between the start of treatment and death directly due to the disease.
Effects on pain score in subjects | up to 96 weeks
  Questionnaire: pain score：The line segments below all have numbers from 0 to 10, where 0 means no pain and 10 is the worst pain you can imagine.
Effects on subjects' health-related quality of life | up to 96 weeks
  Questionnaire: Quality of life related scale（The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 3rd edition）.For questions 1 to 28, choose a number from 1 to 4. 1 means none and 4 means very.For questions 29 and 30, choose a number from 1 to 7, with 1 being very poor and 7 being very good.
Effects on subjects' related symptoms | up to 96 weeks
  Patients' overall impression of severity of cancer symptoms (self-reported)
Effects on pain interference index in subjects | up to 96 weeks
  Questionnaire: pain interference index：Please answer each one by circling a number from 0 to 6, where 0 means none at all and 6 means completely

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital ，Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China